CLINICAL TRIAL: NCT03473015
Title: Oxford Acute Myocardial Infarction - Pressure-controlled Intermittent Coronary Sinus Occlusion
Acronym: OxAMI-PICSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Miracor Medical SA (Industry)
Responsible Party: Principal Investigator, Adrian Banning, Consultant Cardiologist, Professor of Interventional Cardiology, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OxfordRadcliffeH
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-02

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICSO arm (Experimental): STEMI patients with elevated pre-stenting index of microcirculatory resistance (IMR) greater than 40 units treated with pressure-controlled intermittent coronary sinus occlusion (PICSO)
  Interventions: Device: PICSO
- Control (No Intervention): Matched historical cohort of STEMI patients with elevated IMR greater than 40, not treated with PICSO

INTERVENTIONS:
Device: PICSO — The PICSO Impulse catheter is a 8F double lumen catheter with a 15.5x20mm long balloon at the distal end. The balloon inflates and deflates cyclically once deployed in the coronary sinus, leading to intermitted coronary sinus pressure increase. The catheter is connected to the console through two pneumatic tubes in which helium is shuttled to and from the balloon. In addition, the coronary sinus pressure is monitored through the center lumen of the catheter.
  Arms: PICSO arm

SUMMARY:
The OxAMI-PICSO is a study about the use of pressure controlled intermittent coronary sinus occlusion (PICSO) to improve the treatment of patients presenting with heart attack. PICSO is a device consisting of a balloon which is deployed in the coronary sinus. When inflated the balloon can improve the blood flow to the region of heart affected by the heart attack. The study aims to analyse the potential benefit of PICSO in improving blood flow to heart muscle in a selected group of patients admitted with a large heart attack involving the anterior wall of the heart. The comparator group will be a well-matched group of participants of the ongoing OxAMI study.

In order to select patients with a large heart attack, we will measure the index of microcirculatory resistance (IMR), before completion of the heart attack treatment procedure. The IMR value provides measurement of the blood flow at the level of the tiny vessels branching from the large coronary arteries. Our preliminary data from the OxAMI study have shown that an IMR > 40 suggests that the patient is having a large myocardial infarction (heart attack). Only patients with starting IMR > 40 will be considered eligible for the PICSO treatment.

The benefit of PICSO will be assessed by measuring 1) indexes of coronary blood flow, 2) the extension of the infarcted area and 3) the levels of different molecules released in the blood.

DETAILED DESCRIPTION:
The OxAMI-PICSO study is a prospective single centre observational cohort study of the use of pressure-control intermittent coronary sinus occlusion (PICSO) in patients presenting for primary percutaneous coronary intervention (PCI) for acute myocardial infarction.

Patients, age 30-90, presenting with ST elevation myocardial infarction will be considered for inclusion in the study. Measurement of index of microcirculatory resistance (IMR) before stenting is an essential prerequisite for the study: only patients with pre-stenting IMR > 40 will be considered eligible for the PICSO treatment. Patients with IMR≤ 40 will remain in the study but will not undergo PICSO treatment.

The procedure for consent in patients undergoing emergency PCI will be as already established in the ongoing OxAMI study (Ethics Ref 11/SC/0397) Because of the urgency of the situation it is not feasible to obtain fully informed written consent. Fully informed consent requires that the potential participant have time to read and reflect on a patient information sheet which in this context is clinically inadvisable. We therefore propose to obtain verbal assent so as to optimize the amount of appropriate information conveyed to potential participants acutely and minimize the clinical risks involved with substantial delay. The research study will be discussed verbally with the patient and the risks and benefits explained. Only conscious patients, able to provide verbal assent will be enrolled in the study.

In detail the patient at the time of verbal assent process will be informed that as part of the research project he/she might undergo to measurement of the index of microcirculatory resistance (IMR) which allows to have an indirect assessment of the entity of the ongoing heart attack. The patient will be also informed that in case IMR value will be greater than 40, thus suggesting a possible significant damage to the heart muscle that may benefit from additional treatment, he/she might be asked to provide assent for PICSO treatment. Patients with pre-stenting IMR ≤ 40 or those with pre-stenting IMR > 40 who elect not to receive PICSO treatment will be given the opportunity to continue to participate within the OxAMI-PICSO study, but without the use of the PICSO device.

Participants will be reminded that they have the right to withdraw from the study at any stage and that this will not affect their treatment or human rights. Once the emergency phase is over and treatment has been delivered, full written informed consent will be sought as soon as practical. For most patients this means within 12 hours of admission.

The PCI procedure will be undertaken in a standard fashion, and include the use of pressure wire measurements before and after stent deployment.

Only patients with pre-stenting IMR > 40 and who assent to receive PICSO treatment will undergo 24 hours coronary angiogram with coronary physiology measurement, 24-48 hours CMR scan and 6 months CMR scan. Patients who assent to participate in the study but in whom the pre-stenting IMR ≤ 40, or those in whom the pre-stenting IMR > 40 but the participant declines PICSO treatment will remain in the study for clinical data collection only at the same follow up time points (24 hours, 48 hours and 6 months).

The control group of the OxAMI-PICSO study will be represented by a matched cohort of patients with STEMI with pre-stenting IMR greater than 40 units already enrolled as part of the OxAMI study (Ethics Ref 11/SC/0397)

In details the OxAMI-PICSO study will consist of five stages:

Stage 1: Pre-Stenting

1. Diagnostic angiography will be performed in the standard manner using appropriate catheters.
2. Bivalirudin will be administered (0.75mg/kg bolus followed by an infusion of 1.75 mg/kg/min for up 4 hours after the procedure as clinically warranted), as routinely used for PCI. The lesion will be crossed with a coronary guide wire in the usual manner for PCI. Normal blood flow will be rapidly achieved by thrombus aspiration and/or predilation
3. Pre-stenting IMR will be measured, using a pressure wire, as used for routine clinical measurements in patients undergoing PCI.
4. If pre-stenting IMR is > 40, patients will be invited to receive the PICSO device. If pre-stenting IMR is ≤ 40 PICSO device will not be proposed, but the patient will be invited to remain in the study for routine clinical data collection.

Stage 2: PICSO treatment

1. In patients with IMR >40 who assent to PICSO treatment, the PICSO device will be deployed and PICSO treatment delivered until a PICSO dose of 800 mmHg is achieved

Stage 3: Stenting

1. Stenting is performed as usual clinical practice.
2. Post-dilation is left to operator's discretion, as in clinical routine.
3. At the end of the procedure a final reassessment of IMR is performed again as previously described.

Stage 4: 24-48 hours post PCI

Full written consent to take part to the OxAMI-PICSO study is obtained as soon as practicable. The following study assessments may be carried out:

1. Repeat coronary angiogram for assessment of coronary physiology parameters assessment - for participants who receive the PICSO device only
2. Cardiac magnetic resonance - for participants who receive the PICSO device only
3. Data Collection, Patient Reported Outcomes and Cardiovascular Outcomes

Stage 5: 6 months post PCI Participants will be invited to attend the hospital as an outpatient at approximately 6 months post-PPCI for the following research assessments

1. Cardiovascular MRI - for participants who receive the PICSO device only
2. Data Collection, Patient Reported Outcomes and Cardiovascular Outcomes

Recruitment to the study will cease as soon as 25 participants have undergone PICSO treatment and have completed follow-up at 6 months. The study will end on the date of the last CMR at 6 months follow up of the last participant recruited.

Sample Size

The OxAMI-PICSO study aims to investigate the potential benefit of PICSO in a highly selected population of STEMI patients. In line with the data reported by Sayeed et al in a previous metanalysis on 7 studies about PICSO application in animal models, the recently published Prepare-RAMSES study also observed a 30% reduction in IS in the treatment arm, however such reduction was not statistically significant in comparison to the control arm. The study, however could still show a benefit of PICSO in terms of IS reduction at six months follow up in the subgroup of patients receiving high PICSO quantity. The study, however, was significantly hampered by the inclusion of relative low risk patients and by a small sample size. The author managed indeed to deliver full PICSO treatment only in 63% of the initial planned cohort (12 patients, of the 30 planned, received a prolonged treatment with PICSO).

In order to address the first limitation of the Prepare-RAMSES study, OxAMI-PICSO study will select patients with a pre-stenting higher IMR. In this way PICSO is meant to be applied only in a population at higher risk and highly likely to get benefit from its application.

In this regard assuming that the stricter inclusion criteria may allow to detect a substantial benefit from PICSO compared to the control group and expecting that this will allow to achieve a significant 29% reduction in IS as shown in Sayeed's metanalysis, we initially calculated a final sample size of 12 patients with complete final data per each group with an interval of confidence at 95% and a 80% power. However, considering that this was the final same sample size enrolled in the Prepare-RAMSES study, initially meant to recruit 30 patients per arm, we propose to double the actual sample size from 12 to 25 per arm.

Allowing for participants who do not wish to undergo repeat cardiac catheterisation, or cardiac MRI, we anticipate that approximately 75 patients may be recruited to the study in order to achieve full participation and complete follow up in 25 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 30 to 90 years,
* Clinical presentation with STEMI
* Referred for coronary angiography with view to proceed to PCI with stenting.

Exclusion Criteria:

* Patients in whom safety or clinical concerns preclude participation.
* Known anaemia (Hb <9).
* Pregnant or breast feeding females.
* Revascularization by mean of balloon angioplasty without stenting
* History of stroke, TIA or reversible ischemic neurological disease within last 6 months
* Known severe renal failure (eGFR < 30 ml/min/1.73m2) or history of dialysis or renal transplant
* Previous coronary bypass artery grafting
* Known severe valvular abnormalities
* Previous STEMI presentation
* Presentation with cardiogenic shock
* Severe bradycardia (Heart rate < 50 beats per minutes)
* STEMI due to stent thrombosis
* Unconscious on presentation
* Non-cardiac comorbidities and life expectancy < 1 year
* Use of warfarin
* Presence of pacemaker or other electrodes in the coronary sinus
* Contraindications to adenosine
* Additional exclusion criteria for participants undergoing CMR

  * claustrophobia which limits / prevents participants from remaining in CMR scanner.
  * patients who cannot lie flat on the scan table.
  * patients with metallic implants, pacemakers, implantable defibrillators etc, unless known to be CMR compatible.
  * patients with known allergy to medium of contrast (gadolinium)

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Banning, MD, MBBS, Study Chair — Adrian.Banning@ouh.nhs.uk
Locations (1):
- Heart Centre - John Radcliffe Hospital - Oxford University Hospitals - NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] De Maria GL, Patel N, Kassimis G, Banning AP. Spontaneous and procedural plaque embolisation in native coronary arteries: pathophysiology, diagnosis, and prevention. Scientifica (Cairo). 2013;2013:364247. doi: 10.1155/2013/364247. Epub 2013 Dec 19. PMID 24455430
- [Background] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, Ho MY, Kim HS, Loh JP, Oldroyd KG. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41. doi: 10.1161/CIRCULATIONAHA.112.000298. Epub 2013 May 16. PMID 23681066
- [Background] De Maria GL, Cuculi F, Patel N, Dawkins S, Fahrni G, Kassimis G, Choudhury RP, Forfar JC, Prendergast BD, Channon KM, Kharbanda RK, Banning AP. How does coronary stent implantation impact on the status of the microcirculation during primary percutaneous coronary intervention in patients with ST-elevation myocardial infarction? Eur Heart J. 2015 Dec 1;36(45):3165-77. doi: 10.1093/eurheartj/ehv353. Epub 2015 Aug 7. PMID 26254178
- [Background] De Maria GL, Kassimis G, Raina T, Banning AP. Reconsidering the back door approach by targeting the coronary sinus in ischaemic heart disease. Heart. 2016 Aug 15;102(16):1263-9. doi: 10.1136/heartjnl-2016-309642. Epub 2016 Jun 10. PMID 27288281
- [Background] Mohl W, Mina S, Milasinovic D, Kasahara H, Wei S, Maurer G. Is activation of coronary venous cells the key to cardiac regeneration? Nat Clin Pract Cardiovasc Med. 2008 Sep;5(9):528-30. doi: 10.1038/ncpcardio1298. No abstract available. PMID 18679384
- [Background] Khattab AA, Stieger S, Kamat PJ, Vandenberghe S, Bongoni A, Stone GW, Seiler C, Meier B, Hess OM, Rieben R. Effect of pressure-controlled intermittent coronary sinus occlusion (PICSO) on myocardial ischaemia and reperfusion in a closed-chest porcine model. EuroIntervention. 2013 Jul;9(3):398-406. doi: 10.4244/EIJV9I3A63. PMID 23872654
- [Background] Syeda B, Schukro C, Heinze G, Modaressi K, Glogar D, Maurer G, Mohl W. The salvage potential of coronary sinus interventions: meta-analysis and pathophysiologic consequences. J Thorac Cardiovasc Surg. 2004 Jun;127(6):1703-12. doi: 10.1016/j.jtcvs.2004.01.036. PMID 15173727
- [Background] Mohl W, Glogar DH, Mayr H, Losert U, Sochor H, Pachinger O, Kaindl F, Wolner E. Reduction of infarct size induced by pressure-controlled intermittent coronary sinus occlusion. Am J Cardiol. 1984 Mar 15;53(7):923-8. doi: 10.1016/0002-9149(84)90526-5. PMID 6702648
- [Background] Van de Hoef TP, Nolte F, Delewi R, Henriques JP, Spaan JA, Tijssen JG, Siebes M, Wykrzykowska JJ, Stone GW, Piek JJ. Intracoronary hemodynamic effects of pressure-controlled intermittent coronary sinus occlusion (PICSO): results from the First-In-Man Prepare PICSO Study. J Interv Cardiol. 2012 Dec;25(6):549-56. doi: 10.1111/j.1540-8183.2012.00768.x. Epub 2012 Sep 20. PMID 22994798
- [Background] van de Hoef TP, Nijveldt R, van der Ent M, Neunteufl T, Meuwissen M, Khattab A, Berger R, Kuijt WJ, Wykrzykowska J, Tijssen JG, van Rossum AC, Stone GW, Piek JJ. Pressure-controlled intermittent coronary sinus occlusion (PICSO) in acute ST-segment elevation myocardial infarction: results of the Prepare RAMSES safety and feasibility study. EuroIntervention. 2015 May;11(1):37-44. doi: 10.4244/EIJY15M03_10. PMID 25868741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: OxAMI-PICSO is a single-centre, investigator-initiated study, prospectively enrolling patients with anterior STEMI admitted for pPCI at the Oxford Heart Centre from July 2015 to September 2017.
Pre-assignment Details: Patients with pre-stenting IMR ≤40 units and patients with an IMR >40 unwilling to be treated with PICSO or in case of PICSO unavailability were enrolled in the parallel running observational Oxford Acute Myocardial Infarction (OxAMI) study (REC 10/H0408/24)2.
  Between December 2015-September 2016, OxAMI-PICSO was paused due to an expired CE mark on the device, requiring a new submission to the local ethics committee for approval, which ultimately allowed resumption of recruitment.
Groups:
- PICSO Treatment Group: STEMI patients with elevated pre-stenting index of microcirculatory resistance (IMR) greater than 40 units treated with pressure-controlled intermittent coronary sinus occlusion (PICSO)
  PICSO: The PICSO Impulse catheter is a 8F double lumen catheter with a 15.5x20mm long balloon at the distal end. The balloon inflates and deflates cyclically once deployed in the coronary sinus, leading to intermitted coronary sinus pressure increase. The catheter is connected to the console through two pneumatic tubes in which helium is shuttled to and from the balloon. In addition, the coronary sinus pressure is monitored through the center lumen of the catheter.
- Pre-stenting IMR ≤ 40 Group: STEMI patients with pre-stenting index of microcirculatory resistance (IMR) equal or less than 40 units not treated with pressure-controlled intermittent coronary sinus occlusion (PICSO)
- Control Group: Matched historical cohort of STEMI patients with elevated IMR greater than 40, not treated with PICSO
Period: Overall Study
Arm/Group | PICSO Treatment Group | Pre-stenting IMR ≤ 40 Group | Control Group
Started | 25 | 30 | 50
Post-stenting IMR | 25 | 30 | 50
IMR Reassessment 24-48 Hours Post-PCI | 20 | 0 (IMR was not reassessed in this group as the pre-stent IMR was equal or less than 40 units) | 31
Acute Cardiac MRI Within 24 Hours | 17 | 17 | 29
Cardiac MRI at 6 Months | 14 | 16 | 24
Completed | 25 | 30 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-stenting IMR ≤ 40 Units Group: STEMI patients with pre-stenting index of microcirculatory resistance (IMR) equal or less than 40 units not treated with pressure-controlled intermittent coronary sinus occlusion (PICSO)
- Total: Total of all reporting groups
Arm/Group | PICSO Treatment Group | Pre-stenting IMR ≤ 40 Units Group | Control Group | Total
Number analyzed (Participants) | 25 | 30 | 50 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] — Variables reported as Mean (Standard Deviation)
  years | 65.6 (10.9) | 59.6 (9.4) | 60.4 (10.2) | 61.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants
    Female | 6 | 6 | 7 | 19
    Male | 19 | 24 | 43 | 86
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 25 | 30 | 50 | 105
Hypertension [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants | 12 | 15 | 22 | 49
Hypercholesterolaemia [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants | 4 | 11 | 15 | 30
Active smoker [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants | 9 | 13 | 23 | 45
Diabetes [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants | 6 | 3 | 14 | 23
Family history of coronary artery disease [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants | 8 | 11 | 23 | 42
Previous history of coronary artery disease [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants | 3 | 5 | 15 | 23
Ischaemic time [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants
    <3 hours | 15 | 19 | 20 | 54
    ≥ 3 hours and <6 hours | 5 | 11 | 15 | 31
    ≥ 6 hours | 5 | 0 | 15 | 20
Number vessel disease [Count of Participants; unit: Participants] — Frequencies (Percentage%)
  Participants
    1 vessel disease | 19 | 24 | 35 | 78
    2 vessel disease | 6 | 3 | 8 | 17
    3 vessel disease | 0 | 3 | 7 | 10
Thrombolysis in myocardial infarction (TIMI) flow at presentation [Count of Participants; unit: Participants] — Patients were graded as follow TIMI 0 = no antegrade flow beyond the point of occlusion. TIMI 1= contrast dye passes beyond the obstruction but fails to opacify the entire coronary bed distal to the obstruction TIMI 2= contrast dye passes across the obstruction and opacifies the coronary bed distal to the obstruction. The rate of entry and clearance of the contrast material into the vessel is slower compared to non-infarcted related vessel TIMI 3= normal antegrade flow, entry and clearance of contrast dye similar as in non-infarct related artery
  Lower TIMI flow = worse outcome
  Participants
    0 | 22 | 21 | 43 | 86
    1 | 1 | 2 | 2 | 5
    2 | 2 | 2 | 4 | 8
    3 | 0 | 5 | 1 | 6
Angio-thrombus score [Count of Participants; unit: Participants] — Angio-Thrombus Score 0 = no thrombus Angio-Thrombus Score 1= possible thrombus Angio-Thrombus Score 2= thrombus length <1/2 vessel diameter Angio-Thrombus Score 3 = thrombus length > 1/2, but < 2 vessel diameter Angio=Thrombus Score 4 = thrombus length <1/2 vessel diameter Angio Thrombus Score 5 = vessel still occluded after passage of guide wire
  Higher Thrombus Score = worse outcome
  Participants
    0-1-2 | 1 | 4 | 7 | 12
    3 | 1 | 9 | 10 | 20
    4 | 12 | 11 | 23 | 46
    5 | 11 | 6 | 10 | 27
Age thrombus burden index of Microcirculatory Resistance (ATI) score [Count of Participants; unit: Participants] — ATI Score can range from 0 to 6 (the higher the worse) and is calculated by adding points given to each of the following variables
  Age < 50 years = 0 point > 50 years = 1 point
  Angio Thrombus Score 0-3 = 0 point 4 = 1 point 5 = 3 points
  Index of Microcirculatory resistance (IMR) < 40 U = 0 point 40 U - 100 U = 1 point > 100 U = 2 points
  Participants
    0-1 | 0 | 16 | 4 | 20
    2-3 | 12 | 10 | 33 | 55
    4-5-6 | 13 | 4 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: Index of Microcirculatory Resistance
Description: Assessment of coronary microvascular status using IMR
  IMR is calculated as the product of distal coronary pressure and transit time of bolus of saline during hyperaemic condition. It is a continuous variable that can range from to infinite value. Despite technically it represents a product of pressure in mmHg and time (seconds), by convention it is expressed in Units. A normal IMR value is accepted to be < 25 U, however in STEMI patients (as in the cohort reported in the study) an IMR > 40 U is associated to worse clinical outcome
Time Frame: 48 hours post primary percutaneous coronary intervention
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | PICSO Treatment Group | Control Group
Number analyzed (Participants) | 20 | 31
units | 24.8 [18.5 to 35.9] | 45.0 [32.0 to 51.3]

2. Secondary Outcome: Infarct Size
Description: Infarct size measured by Cardiac magnetic resonance
  Infarct size is measured at cardiac magnetic resonance imaging scan and is expressed as hyperhanced core after gadolinium contrast dye injection. Infarct size is measured in gram of myocardial tissue and for standardization typically expressed and reported as percentage of whole left ventricular myocardial mass.
Time Frame: 24-48 hours post primary percutaneous coronary intervention
Measure: Median (Inter-Quartile Range); unit: percentage of left ventricular mass
Arm/Group | Pre-stenting IMR ≤ 40 Units Group | Control Group | PICSO Treatment Group
Number analyzed (Participants) | 17 | 29 | 17
percentage of left ventricular mass | 23.0 [19.0 to 53.9] | 41.0 [31.5 to 46.0] | 39.0 [27.5 to 44.0]

3. Secondary Outcome: Infarct Size 6 Months
Description: as for outcome 2
Time Frame: 6 months post primary percutaneous coronary intervention
Measure: Median (Inter-Quartile Range); unit: percentage of left ventricular mass
Arm/Group | Pre-stenting IMR ≤ 40 Units Group | Control Group | PICSO Treatment Group
Number analyzed (Participants) | 16 | 24 | 14
percentage of left ventricular mass | 19.0 [10.7 to 28.0] | 33.0 [28.0 to 37.0] | 26.0 [20.2 to 30.0]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pre-stenting IMR ≤ 40 Units Group | Control Group | PICSO Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/50 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 0/30 | 0/50 | 0/25

LIMITATIONS AND CAVEATS:
OxAMI-PICSO was a non-randomised study. Another limitation is the number of patients without cardiac MRI (cMRI). This is a common finding in an emergency all-comers design but, while cMRI within 24-48 hours was performed in only 60% of the study population, most of these patients completed follow-up with cMRI at six months (85.7%). Thirdly, the ATI score was not used to select high-risk STEMI patients, since it was not yet validated at the time of study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT03473015/Prot_SAP_000.pdf